CLINICAL TRIAL: NCT05008848
Title: Reaching Rural Cancer Survivors Who Smoke Using Text-Based Cessation Interventions
Brief Title: Reaching Rural Cancer Survivors Who Smoke Using Text-Based Program
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A211901; NCI-2021-03543 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH)
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Health Promotion; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (SGR program, text messages) (Experimental): Patients participate in schedule gradual reduction program over 8 weeks to reduce the frequency of cigarette use. Patients also receive cessation support messages via text messages for 12 weeks.
  Interventions: Behavioral: Smoking Cessation Intervention; Other: Health Promotion and Education; Other: Questionnaire Administration
- Group II (booklet) (Active Comparator): Patients receive NCI's Clearing the Air booklet to help plan to gradually quit smoking.
  Interventions: Other: Informational Intervention

INTERVENTIONS:
Behavioral: Smoking Cessation Intervention — Participate in schedule gradual reduction program
  Arms: Group I (SGR program, text messages)
Other: Health Promotion and Education — Receive cessation support messages
  Arms: Group I (SGR program, text messages)
Other: Informational Intervention — Receive NCI's Clearing the Air booklet
  Arms: Group II (booklet)
Other: Questionnaire Administration — Ancillary studies
  Arms: Group I (SGR program, text messages)

SUMMARY:
This phase III trial compares the effect of text-based cessation intervention to a manual in helping rural cancer patients who smoke, quit. Text-based scheduled gradual reduction may reduce the frequency of cigarette use to zero and may be effective in quitting smoking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of an eight-week text-based scheduled gradual reduction (SGR) intervention (a personalized eight-week reduction schedule paired with National Cancer Institute's [NCI's] Smokefree.TXT) compared to a control intervention (NCI Clearing the Air Cessation Booklet) on biochemically-validated smoking cessation six-month post-quit date in rural cancer survivors.

SECONDARY OBJECTIVE:

I. Compare the efficacy of the eight-week text-based SGR intervention and a control intervention on Linear Analog Self-Assessment (LASA)-6 overall quality of life (QOL) at 30-days post-quit date and six-months post-quit date.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients participate in schedule gradual reduction program over 8 weeks to reduce the frequency of cigarette use. Patients also receive cessation support messages via text messages for 12 weeks.

GROUP II: Patients receive NCI's Clearing the Air booklet to help plan to gradually quit smoking.

After completion of study, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a cancer diagnosis within the past 10 years, and can currently be receiving curative treatment
* Not currently on hospice
* Currently smokes >= 5 cigarettes daily
* Lives in a nonmetro/rural county (defined as having a Rural Urban Continuum Code [RUCC] code of 4-9)
* Patient interested in participating in a smoking cessation program, and not currently participating in a smoking cessation clinical trial
* Not currently using any smoking cessation pharmacotherapy (e.g. nicotine replacement therapy, bupropion or varenicline), or currently participating in any cessation program
* Patient has a cell phone or smart phone device with texting ability
* In order to complete the mandatory patient-completed measures, participants must be able to speak and read English
* Age >= 18 years
* Participant must be willing to provide a urine sample.

Exclusion Criteria:

* Psychiatric illness which would prevent the patient from giving informed consent
* Patients with impaired decision-making capacity are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2028-03-26 (Estimated); Study Completion 2028-08-26 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated tobacco cessation | Up to 6 months post-quit date
  Response will be defined as (1) urine cotinine levels < 50 ng/ml or (2) urine cotinine levels >=50 ng/ml and an urine anabasine level < 2 ng/ml if a patient self-reports vaping use or the use of nicotine replacement therapy (NRT). Patients who do not return at 6 months post-quit date for the cotinine assessment (and anabasine, if applicable) will be deemed non-responders. The analysis population is defined as all randomized and eligible patients. The primary evaluation of the primary outcome will be the covariate-adjusted intervention effect (adjusted odds ratio) obtained from a multiple logistic regression model adjusted for the three stratification factors baseline daily cigarette consumption, age, and sex as well as the potential confounding variables cancer diagnosis, cancer type, receipt of chemotherapy, receipt of radiation therapy, and active treatment.

SECONDARY OUTCOMES:
Serially measured overall quality of life (QoL) scores obtained at baseline and at 30-days and 6-months post-quite date | Up to 6-months post-quit date
  At a given measurement time point, the patient-reported overall QoL score will be obtained from a linear analogue self-assessment scale (LASA), which is an 11-point scoring scale (0, 1, …, 10) where 0 indicates as bad as can be and 10 indicates as good as can be. A linear mixed model will be used to compare the average difference between the randomized arms across the two post-randomization time points after adjusting for the baseline overall QoL score, the three stratification factors baseline daily cigarette consumption, age, and sex as well as the potential confounding variables cancer diagnosis, cancer type, receipt of chemotherapy, receipt of radiation therapy, and active treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Devon Noonan, PhD, MPH, FNP-BC, Study Chair — Duke School of Nursing
Locations (207):
- United States (207):
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Saint Helena Hospital, St. Helena, California
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Northeast Georgia Medical Center Braselton, Braselton, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - The Longstreet Clinic - Gainesville, Gainesville, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Carle BroMenn Outpatient Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - HaysMed, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Cancer Center of Acadiana, Lafayette, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Novant Health Colon and Rectal Clinic, Clemmons, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Novant Health Breast Surgery - Greensboro, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Regional Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - STCC at DHR Health Institute for Research and Development, Edinburg, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - Chesapeake Regional Medical Center, Chesapeake, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Sentara Princess Anne Hospital, Virginia Beach, Virginia
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - SSM Health Dean Medical Group - Baraboo, Baraboo, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - SSM Health Dean Medical Group - Janesville, Janesville, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Memorial Hospital of Sweetwater County, Rock Springs, Wyoming

IPD SHARING:
Plan to Share IPD: Yes